CLINICAL TRIAL: NCT03533972
Title: Effect of Ashwagandha (Withania Somnifera) as an Adjunct to Scaling and Root Planing on Salivary Antioxidant and Serum c Reactive Protein Levels in Chronic Generalized Periodontitis- a Randomized Double Blind Clinico-biochemical Trial
Brief Title: Effect of Ashwagandha on Salivary Antioxidant and Serum c Reactive Protein in Chronic Generalized Periodontitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, Dr.Nibha Suneel Kulkarni, Principal Investigator, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: nibhask
Record Dates: First submitted 2018-05-09; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): subjects will be provided with Ashwagandha capsules 500 mg twice daily, after meals with plain water for 1 month
  Interventions: Drug: Ashwagandha
- Control group (Placebo Comparator): subjects will be provided with placebo capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ashwagandha — ashwagandha capsules given to the subjects twice daily after meals for 1 month
  Other Names: withania somnifera
  Arms: Test group
Other: Placebo — placebo capsules given twice daily after meals for 1 month
  Arms: Control group

SUMMARY:
Periodontal disease is an immune-inflammatory disease which consists of connective tissue breakdown, loss of attachment, and alveolar bone loss.In normal physiology, there is an equilibrium maintained between reactive oxygen species (ROS) activity and antioxidant defence capacity. when this equilibrium changes and shifts in favour of ROS, it will result in oxidative stress (OS). Increased levels of acute phase proteins have been associated with gingival inflammation and periodontitis, which reflected the locally stressed environment. it has been well established that in chronic inflammation sites there is over-production of ROS. The human body consists of an array of antioxidant defense mechanisms (non-enzymatic and enzymatic antioxidants) which removes harmful ROS as soon as they are formed and prevent their deleterious effects. Superoxide dismutase (SOD), catalase (CAT), and glutathione peroxidase are the enzymatic antioxidants, while the nonenzymatic antioxidants include vitamins E and C, and reduced glutathione. C - reactive protein (CRP) is a plasma protein that reflects a measure of the acute phase response to inflammation and is one of the markers of choice in monitoring this response. Changes in peripheral blood cellular and molecular components can be seen in patients with periodontitis, as periodontitis includes inflammatory changes of the periodontal tissues. Ashwagandha is also known as Indian ginseng and winter cherry. It consists of dried roots of Withania Somnifera (Family: Solanaceae).6 The Sanskrit words ashva meaning horse, and gandha meaning smell together form the name Ashwagandha. Ashwagandha possessed marked anti-inflammatory effect against denaturation of protein in vitro. the effect was plausibly due to the alkaloid and withanolide contents of ashwagandha. It is a multipurpose herb, which acts as adaptogenic, antioxidant, anticancer, anxiolytic, antidepressant, cardio protective, thyroid modulating, immunomodulating, antibacterial, anti-inflammatory, neuroprotective, cognitive enhancing and hematopoietic agent.So, this study is carried out to assess SOD & CRP levels with or without Ashwagandha supplementation as an adjunct to scaling and root planing(SRP) in chronic periodontitis(CP) patients.

DETAILED DESCRIPTION:
Periodontal disease is an immune-inflammatory disease which consists of connective tissue breakdown, loss of attachment, and alveolar bone loss.1 In normal physiology, there is an equilibrium maintained between reactive oxygen species (ROS) activity and antioxidant defence capacity. Thus when this equilibrium changes and shifts in favour of ROS, it will result in oxidative stress (OS). OS plays a causative role in pathogenesis of periodontal disease.2 Increased levels of acute phase proteins have been associated with gingival inflammation and periodontitis, which reflected the locally stressed environment.3 The human body consists of an array of antioxidant defense mechanisms (non-enzymatic and enzymatic antioxidants) which removes harmful ROS as soon as they are formed and prevent their deleterious effects. Superoxide dismutase (SOD), catalase (CAT), and glutathione peroxidase are the enzymatic antioxidants, while the nonenzymatic antioxidants include vitamins E and C, and reduced glutathione.2 C - reactive protein (CRP) is a plasma protein that reflects a measure of the acute phase response to inflammation and is one of the markers of choice in monitoring this response. CRP can be used for the prediction and early detection of periodontal disease as it is a sensitive marker to evaluate the inflammatory status.4 Ayurveda is the traditional system of medicine practiced in India that can be traced back to 6000 BC .It is a basic foundation of ancient medical science in India. Ashwagandha is also known as Indian ginseng and winter cherry. It consists of dried roots of Withania Somnifera (Family: Solanaceae).6 The Sanskrit words ashva meaning horse, and gandha meaning smell together form the name Ashwagandha. The root has been described as having a strong "horse like" aroma, although some experts note that the origin of the name suggests that one who ingests it can attain the strength and vitality of a horse.7 Ashwagandha possessed marked anti-inflammatory effect against denaturation of protein in vitro. the effect was plausibly due to the alkaloid and withanolide contents of ashwagandha.6 Ashwagandha root has major bioactive constituents which are steroidal alkaloids and lactones known as withanolides which have immunomodulatory effect.8 It is a multipurpose herb, which acts as adaptogenic, antioxidant, anticancer, anxiolytic, antidepressant, cardio protective, thyroid modulating, immunomodulating, antibacterial, antifungal, anti-inflammatory, neuroprotective, cognitive enhancing and hematopoietic agent.7 Also, by taking Ashwagandha regularly one can enhance his memory and learning skills dramatically.9So, this study is carried out to assess SOD & CRP levels with or without Ashwagandha supplementation as an adjunct to scaling and root planing(SRP) in chronic periodontitis(CP) patients.

MATERIALS AND METHODS

The study will be a randomized double-blind clinical and biochemical trial in which 50 subjects with CP in the age group of 30-55 years, reporting to Department of Periodontology, TKDC and RC, New Pargaon will be equally and randomly divided into Test Group (TG) and Control Group (CG). The randomization will be done based on consort guidelines 2010 14

TG will be provided with Ashwagandha capsules 500 mg twice daily, after meals with plain water for 1 month and CG will be provided with placebo. SRP will be done at baseline in TG and CG. Clinical and biochemical parameters will be recorded at baseline, 1st month (4 weeks) and 2nd month (8 weeks). Whole saliva sample (unstimulated) will be collected. Recall visits will be carried out on 4th week and 8th week. Oral hygiene instructions and reinforcement will be carried out.

Questionnaire will be provided to both the groups for evaluation. All participants will be explained the need and design of the study and written consent will be obtained from each individual prior to the commencement of the study.

Special Instructions Given Regarding with Diet to the Patients during Ashwagandha supplementation period:-

1. No Deep Fry Food should be eaten.
2. No Sour substances.
3. No Pastry Flour (Maida) made foodstuffs.

SAMPLE COLLECTION METHOD-

A ] SALIVA- 2 ml of unstimulated saliva will be collected in a sterile container. Centrifugation will be done for 10 minutes at 4000 rpm.16 Then the supernatant will be removed and stored at 2oC till the assay procedure.

Collection of Saliva Sample: Mahvash Navazesh 200817 Unstimulated whole saliva will be collected for the estimation of SOD.2ml will be collected from each subject between 9.00-10.00a.m.The participants will be requested not to eat or drink anything except water in the morning before sampling. This will ensure that the variability in salivary flow and composition be minimum due to diurnal variation. The subject will be asked to rinse the mouth with distilled water thoroughly to remove any food debris.

B) Serum CRP detection

Samples:

Three ml of venous blood were taken from all patients at baseline, after 4 weeks and 8 weeks.

METHODS OF BIOCHEMICAL ANALYSIS- SOD- Kajridas method C Reactive Protein- hs CRP- Nephelometry.

STATISTICAL ANALYSIS WILL BE DONE BY USING:

With 95% confidence and 80% power minimum 46 patients from either groups, test as well as control group, is required to be included in the study. To compensate for potential dropouts, 50 patients will be considered, 25 patients constituting in each group.

Tests will be done are:-

1. ANOVA repeated measures post hoc.
2. Independent T test.

ELIGIBILITY:
Inclusion Criteria:

* Patients without any known systemic diseases.
* Patients with chronic generalized periodontitis based on CDC 2007

Exclusion Criteria:

* Patients who have taken anti-inflammatory/antibiotic/antioxidant within 3 months of beginning of study.
* Subjects who have undergone periodontal treatment within 6 months of inception of study.
* Tobacco habits in any form and alcoholics.
* Pregnant and lactating women.
* Patients on anti-depressant, thyroid, anti- psychiatric, diabetic medications

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
change in c reactive protein | 1 month and 2 months
  c reactive protein levels by nephelometry
change in super oxide dismutase | 1 month and 2 months
  super oxide dismutase levels by biochemical kazaridas method
change in probing depth | 1 month and 2 months
  measured with UNC 15 Probe
change in clinical attachment loss | 1 month and 2 months
  measured with UNC 15 probe

SECONDARY OUTCOMES:
gingival index | 1 month and 2 months
  clinically assessed its a scale ranging from 0 to 3,in which 0 being the least and 3 being the highest

CONTACTS AND LOCATIONS:
Locations (1):
- Tatyasaheb Kore Dental College, Kolhāpur, Maharashtra, India